CLINICAL TRIAL: NCT02073253
Title: Effect of Noninvasive Ventilation in Thoracic-abdominal Kinematics of Individuals With Heart Failure Associated With Cardiomegaly: a Randomized Controlled Trial
Brief Title: Noninvasive Ventilation and Thoracic-abdominal Kinematics in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Pronto Socorro Cardiológico de Pernambuco-PROCAPE (Unknown)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DissertaçãoLarissaPOE
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without performing any operation (Phase Control) (No Intervention)
- With ventilatory support through NIV (NIV Phase) (Experimental)
  Interventions: Other: Noninvasive ventilation

INTERVENTIONS:
Other: Noninvasive ventilation — In the experimental phase with NIV ventilatory support with bilevel positive pressure was used for 30 minutes with the subject comfortably seated. The NIV (Vivo 40 Bi-Level, General Electric Company) was fitted to the face of volunteer through a face mask, was initially adopted an inspiratory pressure (IPAP) of 15 cm H2O and an expiratory pressure (PEEP) of 5 cmH2O, resulting in a variation in pressure of 10 cm H2O, where the IPAP would be increased, subject to the comfort of the patient until the patient reached a tidal volume of 6-8 ml / kg, not exceeding the maximum of 20 cmH2O for IPAP.
  Arms: With ventilatory support through NIV (NIV Phase)

SUMMARY:
Introduction: Noninvasive ventilation (NIV) has been used to minimize such impairment and increasing ventilator reserve in individuals with heart failure. Aim: To analyze thoracoabdominal kinematics (TK) in individuals with HF associated to cardiomegaly after using NIV. Methods: A randomized crossover clinical trial with allocation consisted of two experimental phases: NIV and control, 7 days apart of each other. During NIV phase, 30 minutes of bi-level ventilation was performed. Any type of ventilator support was offered during control phase. Optoeletronic plethismography was performed to asses TK.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) <30 kg/m2
* functional class II-III according to the New York Heart Association
* of the echocardiogram últiimos 6 months showing ejection fraction (LVEF) ≤ 45%,
* últiimos echocardiogram of six months showing cardiac hypertrophy (left Ventricular Diastolic Diameter (LVDD)> 55mm, Diameter Systolic left Ventricular (LVSD)> 45mm ),
* (optimized from the point of view of drug,
* clinical stability.

Exclusion Criteria:

* unstable angina, myocardial infarction or heart surgery three months before the beginning of the research,
* chronic orthopedic, infectious or metabolic diseases,
* FEV1/FVC <70% predicted characterizing obstructive respiratory disorder;
* active smokers;
* Limitation on the use of NIV: claustrophobia, inability to remain with their mouths closed, abdominal distention, hemodynamic instability, heart rate (HR) <60 bpm, recent trauma, nausea and vomiting face.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Thoraco-abdominal kinematics | Seven days
  The thoraco-abdominal kinematics was performed by optoelectronic plethysmography which were evaluated as primary outcomes: volume change of rib cage (Δv CT), variables related to volume change of rib cage by hemithorax (ΔV ht CT): tidal volume of cash left thoracic (CT VC sx) and tidal volume right ribcage (VC CT dx); variables with distribution volume in different compartments: tidal volume on pulmonary rib cage (VC CTP), tidal volume in abdominal rib cage (VC CTA ) and tidal volume in the abdomen (AB VC).

SECONDARY OUTCOMES:
Other ventilatory responses | Seven days
  The other ventilatory responses were also assessed by optoelectronic plethysmography which were assessed as secondary outcomes: minute ventilation (MV); Inhalant rate (RR), duty cycle (Ti / Ttot), expiratory time (TE), end of rib cage (VEF CT) expiratory volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Fisioterapia da UFPE, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Olson TP, Johnson BD. Influence of cardiomegaly on disordered breathing during exercise in chronic heart failure. Eur J Heart Fail. 2011 Mar;13(3):311-8. doi: 10.1093/eurjhf/hfq177. Epub 2010 Oct 16. PMID 20952768
- See also: database on health — http://www.ncbi.nlm.nih.gov/